CLINICAL TRIAL: NCT05316974
Title: Lymphoedema for Persons With Head- and Neck Cancer
Brief Title: Lymphoedema Among Persons With Head- and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Collaborators: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Eva Ekvall-Hansson, Professor, Lund University
Other Study IDs: 2020-01066
Record Dates: First submitted 2022-03-21; First posted 2022-04-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Cancer of Head and Neck
Keywords: Lymphoedema; Quality of life; Head and neck cancer treatment
MeSH Terms: conditions — Head and Neck Neoplasms; Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Prevalence of lymphoedema — Measures of lymphoedema

SUMMARY:
Lymphedema in the head and neck area is common after treatment for head and neck cancer.

The aim of the research project is:

• to assess the prevalence of lymphedema in patients with head and neck cancer (HNC) by measuring the amount of tissue water in the head and neck area before and after different kinds of cancer treatment, and to evaluate the quality of life before and after cancer treatment.

DETAILED DESCRIPTION:
Measurement of tissue water is performed with a device (MoistureMeterD) see appendix 1. In addition, the neck circumference will be assessed with a measuring tape, according to Purcell (9), see appendix 2. The measurement will be completed by Agneta Hagren, or one of her colleagues, with specific education.

The assessments will be performed before treatment begins as part of the clinical routine (baseline), and at 3 months, and 9 months after treatment completion.

Each participant will respond to quality-of-life QLQ-c30 and QLQ H&N35 questionnaires, appendix 3 and 4, at the same time points as the measurements of tissue water. Ratings of physical activity according to Frändin and Grimby will also be performed (23). The questionnaires will be sent home to the patients before the time for follow-up. A modified LyQLI questionnaire will be given to all patients with lymphedema and filled out at 9 months after treatment completion, appendix 5.

Post-treatment measurements +/- four weeks of the dedicated time point will be considered appropriate.

Discontinuing participation in the trial will be on:

1. Patient request
2. Locoregional tumor progression or failure during the study period. For example, residual neck tumor requiring neck dissection after (C)RT for OPC
3. Locoregional deep infection i.e., suspected abscess at the scheduled time points for measurements.

Any interventional therapy for lymphedema during the follow-up is not cause for exclusion but will be registered.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy or cytology confirmed HNC (all malignant types are accepted) from the oropharynx (OPC), oral cavity (OC) or neck metastases from unknown primary cancer of the head and neck (CUP).
* Tumour stage T1-4, N0-3.
* Planned for treatment with curative intent as recommended at the multidisciplinary tumour board.
* Age >18 years. Able to give informed consent

Exclusion Criteria:

* Previous treatment of HNC or radiation to the head and neck area.
* Planned surgery that includes free tissue transfer or pedicled flaps in the neck (local facial pedicled flaps are accepted).
* Planned neck dissection involving less than three regions of the neck.
* Planned proton therapy.
* Pre-treatment surgery or Botox injections in the tissue in the head and neck area.
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated for head and neck cancer at the ENT department and the Oncology department at Skane University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Change in level of tissue water | Baseline and after 3 and 9 months
  Change in tissue water in the head and neck before and after cancer treatment

SECONDARY OUTCOMES:
QoL | 3 and 9 months
  Quality of life measured by LyQLI
Change in QoL QLQ-c30 | Baseline and after 3 and 9 months
  Change in Quality of life measured by QLQ-c30
Change in QoL QLQ H&N35 | Baseline and after 3 and 9 months
  Change in Quality of life measured by QLQ H&N35
QoL | After 9 months
  Quality of Life measured by Lymphedema Quality of Life Invetory (LyQLI), a scale from

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ekvall Hansson, Professor, Principal Investigator — Lund University, Medical Faculty, Dep of Health Sciences
Locations (1):
- ENT department Skane University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No
According to Swedish law, sharing IPD is not possible. De-identified data can be shared on request